CLINICAL TRIAL: NCT04263701
Title: Effects of Dual Task Training on Gait Parameters in Spastic Diplegic Cerebral Palsy
Brief Title: Dual Task Training in Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Eda Ozge OKUR, Principal Investigator, Kutahya Health Sciences University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMSU
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; dual task training; gait; balance
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Self-controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy Group (Active Comparator): 45 minutes, 2 days in a week for 8 weeks
  Interventions: Other: Therapeutic exercises
- Dual Task Training Group (Experimental): 45 minutes, 2 days in a week for 8 weeks
  Interventions: Other: Dual Task Training

INTERVENTIONS:
Other: Therapeutic exercises — Conventional physiotherapy exercises for children with cerebral palsy
  Arms: Conventional Physiotherapy Group
Other: Dual Task Training — Dual task training in addition to conventional physiotherapy exercises for children with cerebral palsy
  Arms: Dual Task Training Group

SUMMARY:
This study aims to investigate the effects of dual task training on gait and balance parameters, gross motor function skills, functional mobility skills, functional independence levels and health-related quality of life o in children with spastic diplegic cerebral palsy. The clinical study's hypothesis is the dual task training programs are superior to conventional physiotherapy programs to improve the parameters in spastic diplegic cerebral palsy.

DETAILED DESCRIPTION:
In this self-controlled study, children with spastic diplegic cerebral palsy, aged 7-16, who were at level 1 or 2 according to the Gross Motor Function Classification System, scored 27 and above from the Modified Mini Mental Test were included.

Children are recruited to the routine physiotherapy program 45 minutes 2 days a week for 8 weeks, and in addition to the routine physiotherapy program dual task training program 45 minutes 2 days a week for the next 8 weeks. The children will evaluate at baseline, after the routine physiotherapy program and after the dual task training program. Children will be evaluate with Gross Motor Function Measurement-88,Modified Ashworth Scale , gait platform, Edinburgh Visual Gait Score, Pediatric Berg Balance Scale,1 Minute Walk Test, Functional Independence Measure, Pediatric Quality of Life Inventory TM-Cerebral Palsy Module.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with spastic diplegic cerebral palsy,
* Being at level 1 or 2 according to the Gross Motor Function Classification System,
* Being at level 1 according to Communication Function Classification System,
* To adapt to the evaluations,
* To get 27 points or above from the Modified Mini Mental Test (MMMT).

Exclusion Criteria:

* Having had injuries such as strains, sprains or fractures of the lower extremity in the last six months,
* Having undergone a surgical intervention or Botulinum toxin in the last six months,
* Having any known chronic systemic problems,
* Having uncontrollable seizures,
* Having vision or hearing problems.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Gate speed of time-distance gait parameters | Change from baseline time-distance gait parameters at 8th week and 16th week
  Gate speed will be evaluated using with gait platform. The software gives the outcome as km/h.
Step length of time-distance gait parameters | Change from baseline time-distance gait parameters at 8th week and 16th week
  Step lengt will be evaluated using with gait platform. The software gives the outcome as cm and calcules for each lower extremity.
Stride length of time-distance gait parameters | Change from baseline time-distance gait parameters at 8th week and 16th week
  Stride length will be evaluated using with gait platform.The software gives the outcome as cm.
Step time of time-distance gait parameters | Change from baseline time-distance gait parameters at 8th week and 16th week
  Step time will be evaluated using with gait platform.The software gives the outcome as sec and calcules for each lower extremity.
Stride time of time-distance gait parameters | Change from baseline time-distance gait parameters at 8th week and 16th week
  Step time will be evaluated using with gait platform.The software gives the outcome as sec.
Cadance of time-distance gait parameters | Change from baseline time-distance gait parameters at 8th week and 16th week
  Step time will be evaluated using with gait platform.The software gives the outcome as steps/min.
Visual gait analysis | Change from baseline visual gait analysis at 8th week and 16th week
  Visual gait analysis will be performed with Edinburgh Visual Gait Score. Edinburg Visual Gait Score is scoring between 0 to 34 for each lower extremity. The higher scores points above 0 means abnormal gate.
Center of Pressure path length of balance parameters | Change from baseline balance parameters at 8th week and 16th week.
  Center of Pressure path length will be evaluated using with gait platform. The software gives the outcome as mm.
Ellipse area of balance parameters | Change from baseline balance parameters at 8th week and 16th week.
  Ellipse area will be evaluated using with gait platform. The software gives the outcome as mm2.
Functional balance | Change from baseline functional balance at 8th week and 16th week
  Functional balance will be evaluate using with Pediatric Berg Balance Scale. The scale is scoring 0-56. The higher scores indicate better functional balance.

SECONDARY OUTCOMES:
Gross Motor Function Measurement | Change from baseline Gross Motor Function Measurement at 8th week and 16th week
  Gross motor function measurement will be evaluate using with Gross Motor Function Measurement-88. The instrument consist of 5 dimensions which names are A- Lying and rolling, B- Sitting, C- Crawling and Kneeling, D- Standing and E- Walking-running-jumping. Each dimension is scoring 0-100. The higher scores indicate better motor function.
Muscle Tonus | Change from baseline Muscle Tonus at 8th week and 16th week
  Muscle tonus will be evaluate using with Modified Ashworth Scale. This assesment will be performed by a physiotherapist. The Physiotherapist evaluate the muscle tonus of upper and lower extremity muscules. Scoring is between 0-4 and higher scores indicate hypertonus.
Functional Mobility Skills | Change from baseline Functional Mobility Skills at 8th week and 16th week
  Functional mobility skills will be evaluate using with 1-Minute Walk Test. The test perform on a 20 meters platform. The patient walk on the platform as quick as in 1 munite. The walking distance is recorded.
Functional Independence Levels | Change from baseline Functional Independence Levels at 8th week and 16th week
  Functional independence levels will be evaluate using with Functional Independence Measurement (WeeFIM). WeeFIM is consist of 6 part, 18 items. It consists of self-care, sphincter control, locomotion, transfers, communication and social cognition subtitles. Scoring is between 18 to 126 and the higher scores indicate better functional indepence levels.
Health-related quality of life | Change from baseline health-related quality of life at 8th week and 16th week
  Health-related quality of life will be evaluate using with Pediatric Quality of Life Inventory TM. The inventory include daily activities, school activities, movement and balance, pain and hurt, fatique, eating activities and speech and communication subtitles. Each subtitles is scoring 0 to 100 and the higher scores indicate lower problems.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Ozge Okur, Msc, Principal Investigator — KMSU
Locations (1):
- KMSU, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study aims to investigate the effects of dual task training on gait and balance parameters, gross motor function skills, functional mobility skills, functional independence levels and health-related quality of life o in children with spastic diplegic cerebral palsy. The clinical study's hypothesis is the dual task training programs are superior to conventional physiotherapy programs to improve the parameters in spastic diplegic cerebral palsy.

REFERENCES:
- [Derived] Okur EO, Arik MI, Okur I, Gokpinar HH, Gunel MK. Dual-task training effect on gait parameters in children with spastic diplegic cerebral palsy: Preliminary results of a self-controlled study. Gait Posture. 2022 May;94:45-50. doi: 10.1016/j.gaitpost.2022.02.020. Epub 2022 Feb 17. PMID 35247824